CLINICAL TRIAL: NCT00848224
Title: Improving Adherence to Pharmacological Treatment
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Ira S. Ockene, M.D., University of Massachusetts Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HL66786
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Medication Adherence
Keywords: coronary heart disease; lipid lowering medication; NCEP guidelines
MeSH Terms: conditions — Medication Adherence; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental)
  Interventions: Behavioral: systems-based and pharmacist-mediated program

INTERVENTIONS:
Behavioral: systems-based and pharmacist-mediated program — Patients in the SI were seen by a study pharmacists prior to discharge to establish a relationship with the patient, explain the pharmacist's role in the study, provide education about all discharge medications and a medication card listing all medications and their manner of use, and set the framework for the follow-up telephone calls. Patients received pharmacist-delivered adherence counseling telephone contacts that took place at two weeks following discharge, and at months 1, 3, 6, and 9 oriented towards assisting patients to remain adherent to prescribed lipid-lowering and other medications, and also towards ensuring that all patients were either documented to be at the LDL-C goal, or were assisted to reach the goal by facilitating the scheduling of repeat lipid measurement as needed and providing information, guidelines and prompts to the patient's physician or nurse practitioner.
  Other Names: Patient-centered counseling

SUMMARY:
The overall goal of this study was to implement and evaluate the effects of a systems-based and pharmacist-mediated program designed to improve adherence for patients with known coronary heart disease (CHD) to lipid-lowering pharmacologic therapy and of their physicians/nurse practitioners to the National Cholesterol Education Program Guidelines.

DETAILED DESCRIPTION:
Patients were randomly assigned to a usual care condition which consisted of patients provided with usual care only, or to the Special Intervention (SI) condition. The intervention was implemented and coordinated by pharmacists, who utilized for tracking and communication the Lotus Notes®-based system that was developed for the project.

ELIGIBILITY:
Inclusion Criteria:

* was between 30 and 85 years of age;
* had known CHD, defined as the presence of at least one coronary lesion at coronary angiography of >50%.

Exclusion Criteria:

* was unable or unwilling to give informed consent;
* had a history of intolerance to two or more statin drugs;
* planned to move out of the area within one year of recruitment;
* had a poor prognosis such that life expectancy was thought to be <5 years;
* had a psychiatric illness which limited ability to participate; or
* had no telephone.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2000-09; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome evaluated is the percentage of patients with a serum low-density lipoprotein cholesterol (LDL-C) level <70 mg/dl. | One year

SECONDARY OUTCOMES:
Proportion of prescribed lipid-lowering medication taken by patients as measured by a continuous multiple-interval (CMA) measure of medication availability based on pharmacy records. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ira S Ockene, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States